CLINICAL TRIAL: NCT04669561
Title: The Chronology of Lifitegrast Effect on Anterior Surface Rehabilitation (CLEAR) Study: An Investigation on Lifitegrast's Speed of Onset in Improving Ocular Surface Health in Dry Eye Patients
Brief Title: The Chronology of Lifitegrast Effect on Anterior Surface Rehabilitation (CLEAR) Study
Acronym: CLEAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Research Insight LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIF606A1US08T
Record Dates: First submitted 2020-12-09; First posted 2020-12-17 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — lifitegrast; Ophthalmic Solutions

STUDY DESIGN:
Intervention Model Description: This is a multicenter, prospective, open label, self-controlled, single group study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single /arm (Experimental): All patients will receive lifitegrast 5% for 4 weeks and will be evaluated at baseline (before treatment) and at 7, 14, and 28 days.
  Interventions: Drug: Lifitegrast 5% Ophthalmic Solution

INTERVENTIONS:
Drug: Lifitegrast 5% Ophthalmic Solution — Open label, self-controlled, single group study of the efficacy of Lifitegrast 5% in improving higher order aberrations, ocular scatter index, and best corrected visual acuity in patients with dry eye. All patients will receive lifitegrast 5% for 4 weeks and will be evaluated at baseline (before treatment) and at 7, 14, and 28 days.

SUMMARY:
In patients with dry eye, defined as corneal staining and a reduced tear breakup time, lifitegrast will improve higher order aberrations, ocular scatter index, corneal staining, and TBUT as soon as 1 week after initiating treatment.

DETAILED DESCRIPTION:
This is a multicenter, prospective, open label, self-controlled, single group study of the efficacy of Lifitegrast 5% in improving higher order aberrations, ocular scatter index, and best corrected visual acuity in patients with dry eye. All patients will receive lifitegrast 5% for 4 weeks and will be evaluated at baseline (before treatment) and at 7, 14, and 28 days

ELIGIBILITY:
Inclusion Criteria:

* Central or inferior corneal fluorescein staining defined by the Oxford Scale
* Reduced tear break up time (TBUT) ≤ 10 seconds.
* Able to comprehend and sign a statement of informed consent.
* Willing and able to complete all required postoperative visits.

Exclusion Criteria:

* Ocular surgery (e.g., intraocular, oculoplastic, corneal or refractive surgical procedure performed in the study eye within the last 3 months or at any time that in the investigator's clinical judgment if it would interfere with the outcome measures of this study.
* Clinically significant ocular trauma.
* Active ocular Herpes simplex or Herpes Zoster infection
* Ocular inflammation (uveitis, iritis, scleritis, episcleritis, keratitis, conjunctivitis) that is active, at the discretion of the investigator.
* Ocular infection (e.g., viral, bacterial, mycobacterial, protozoan or fungal infection or the cornea, conjunctiva, lacrimal gland, lacrimal sac or eyelids including hordeolum/stye), at the discretion of the investigator.
* Active, systemic or local disease condition that causes clinically significant ocular surface irritation such that it could interfere with the questions in the survey and examination findings, in the opinion of the investigator.
* Moderate to severe (Grade 2-4) allergic, vernal or giant papillary conjunctivitis that would interfere with study findings, in the opinion of the investigator.
* Severe (Grade 3 or 4) inflammation of the eyelid (e.g., blepharochalasis, staphylococcal blepharitis or seborrheic blepharitis)
* Eyelid abnormalities that significantly affect the lid function (e.g., entropion, ectropion, tumor, edema, blepharospasm, lagophthalmos, severe trichiasis, severe ptosis) that would interfere with study findings, in the opinion of the investigator.
* Ocular surface abnormality that may compromise the corneal integrity (e.g., prior chemical burn, recurrent corneal erosion, corneal epithelial defect, Grade 3 corneal fluorescein staining, map dot fingerprint dystrophy, or the effect of any other ophthalmic medication that might in the opinion of the investigator compromise the ocular surface integrity).
* Patients who are under age 18, pregnant or breastfeeding, or who may become pregnant during participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-10-08 (Actual)

PRIMARY OUTCOMES:
Change in corneal higher order aberrations | After 7, 14, and 28 days of treatment.
  Change in corneal higher order aberrations after 7, 14, and 28 days of treatment.

SECONDARY OUTCOMES:
Change in OSI after 7, 14, and 28 days of treatment. | After 7, 14, and 28 days of treatment.
  Change in OSI after 7, 14, and 28 days of treatment.

OTHER OUTCOMES:
Change in best corrected visual acuity after 7, 14, and 28 days of treatment. | After 7, 14, and 28 days of treatment.
  Change in best corrected visual acuity after 7, 14, and 28 days of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: John Hovanesian, MD, Principal Investigator — Research Insight LLC
Locations (3):
- United States (3):
  - Harvard Eye Associates, Laguna Hills, California
  - Bowden Eye & Associates, Jacksonville, Florida
  - Cleveland Eye Clinic, Brecksville, Ohio

IPD SHARING:
Plan to Share IPD: No
The results of the study may be published or presented by the Investigator(s) after the review by, and in consultation and agreement with, the Sponsor, and such that confidential or proprietary information is not disclosed,